CLINICAL TRIAL: NCT02793206
Title: Spectral Domain Optic Cohaerence Tomography Imaging in Patients With Optic Nerve Head Drusen
Brief Title: Spectral Domain OCT Imaging in Patients With Optic Nerve Head Drusen (Tuebingen SD-OCT IN OPTIC NERVE HEAD DRUSEN STUDY)
Acronym: TODS
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 327/2011 BO
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2016-05

CONDITIONS: Optic Disc Drusen
Keywords: Drusen; SD-OCT
MeSH Terms: conditions — Optic Disk Drusen | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Imaging

SUMMARY:
Optic nerve head Drusen are a mostly bilateral change of the optic nerve, eventually causing a slow, but progression loss of the visual fields. Characteristic are the crystalline deposits at the entrance of the optic nerve, the so called optic disc. The material consists of calcium, calcium phosphate, iron, but also amino acids and polysaccharides.

The diagnose is made or confirmed by different imaging modalities like ultrasound and auto-fluorescence imaging. By using the high-resolution imaging with spectral-domain optical coherence imaging (SD-OCT) the volume and deposits at the optic disc can be measured and quantified.

The purpose of this study whether and how defects in the visual fields are related to the deposits. Multimodal imaging of the optic nerve head is planned within the cross-sectional study, at two different time intervals (2 years). Changes in retinal fibre layer (RNFL) thickness and disc parameters are analyzed. Presence and extent of auto-fluorescent changes are evaluated. The prospective trial wants to clarify whether certain parameters at baseline indicate the further outcome and development.

ELIGIBILITY:
Inclusion Criteria:

* patients with Drusen of the optic disc (as proven by ultrasound and clinical appearance)

Exclusion Criteria:

* mental disability
* loss of fixation
* other eye diseases potentially leading to a loss of visual fields

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Optic Disc Drusen
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in RNFL thickness | baseline and 2 years

SECONDARY OUTCOMES:
Loss of Visual Fields | baseline and 2 years
Change in auto-fluorescent areas | baseline and 2 years
Change in Drusen material | baseline and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Asensio-Sanchez VM, Trujillo-Guzman L. SD-OCT to distinguish papilledema from pseudopapilledema. Arch Soc Esp Oftalmol. 2015 Oct;90(10):481-3. doi: 10.1016/j.oftal.2015.05.001. Epub 2015 Jul 3. English, Spanish. PMID 26148443
- [Background] Casado A, Rebolleda G, Guerrero L, Leal M, Contreras I, Oblanca N, Munoz-Negrete FJ. Measurement of retinal nerve fiber layer and macular ganglion cell-inner plexiform layer with spectral-domain optical coherence tomography in patients with optic nerve head drusen. Graefes Arch Clin Exp Ophthalmol. 2014 Oct;252(10):1653-60. doi: 10.1007/s00417-014-2773-5. Epub 2014 Aug 17. PMID 25128962
- [Background] Pilat AV, Proudlock FA, Kumar P, Lee H, Papageorgiou E, Gottlob I. Macular morphology in patients with optic nerve head drusen and optic disc edema. Ophthalmology. 2014 Feb;121(2):552-7. doi: 10.1016/j.ophtha.2013.09.037. Epub 2013 Nov 14. PMID 24238882
- [Background] Sato T, Mrejen S, Spaide RF. Multimodal imaging of optic disc drusen. Am J Ophthalmol. 2013 Aug;156(2):275-282.e1. doi: 10.1016/j.ajo.2013.03.039. Epub 2013 May 12. PMID 23677136